CLINICAL TRIAL: NCT05685745
Title: Multisite Inventory of Neonatal-Perinatal Interventions (MINI) Minimum Dataset
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Nationwide Children's Hospital (Other); University of Iowa (Other); University of Alabama at Birmingham (Other); Jichi Medical University (Other); Saitama Medical University (Other)
Responsible Party: Principal Investigator, Matthew Rysavy, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-22-0578
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-01

CONDITIONS: Infant, Extremely Premature; Obstetric Labor, Premature; Premature Birth; Intensive Care, Neonatal; Intensive Care Units, Neonatal
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the Tiny Baby Collaborative Multicenter Inventory of Neonatal-Perinatal Interventions (MINI) minimum dataset is to serve as a registry detailing the outcomes and practices for all deliveries and infants admitted to intensive care at 22-23 weeks' gestation at participating hospitals.

DETAILED DESCRIPTION:
The minimum dataset collects observational baseline data on both mothers and infants, and the therapies used and outcomes of the infants. The data collected include information on:

* Demographics of mother and infant
* Mother's health, labor and delivery
* Infant's health, medical interventions, and clinical outcomes

These data are used to: provide participating hospitals with reporting for use in quality improvement; evaluate associations between baseline characteristics, treatments, and outcomes; and track trends in disease and therapy.

ELIGIBILITY:
Inclusion Criteria:

* All local births with gestational ages of 22 weeks 0 days - 23 weeks 6 days, regardless of pregnancy outcome or neonatal intensive care (NICU) admission; AND
* All outborn NICU admissions with gestational age at birth of 22 weeks 0 days - 23 weeks 6 days
* Optional: Centers who desire to include data for NICU admissions of infants born <22 weeks' gestation may also submit these data.

Ages: 0 Years to 1 Year | Sex: All
Age Groups: Child
Study Population: Participating hospitals
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Registry of characteristics and outcome data for all deliveries and infants admitted to intensive care at 22-23 weeks' gestation at participating hospitals collected in a uniform manner | Longitudinal database through 1/2028

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Rysavy, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (51):
- United States (37):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Vallywise Health Medical Center, Phoenix, Arizona
  - Miller Children's & Women's Hospital, Long Beach, California
  - Children's Hospital, Orange County, Orange, California
  - University of California, San Diego, San Diego, California
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Wolfson Children's Hospital, Jacksonville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - Orlando Health Winnie Palmer Hospital for Women & Babies, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Grady Memorial, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Nebraska Medicine, Omaha, Nebraska
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Texas Health Resources Harris Hospital, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Women's Hospital of Texas, Houston, Texas
  - CHRISTUS Children's Hospital, San Antonio, Texas
  - Methodist Children's Hospital, San Antonio, Texas
  - St. Luke's Baptist Hospital, San Antonio, Texas
  - North Central Baptist Hospital, San Antonio, Texas
  - Children's Hospital of Richmond, Richmond, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin
- Australia (3):
  - Mater Mother's Hospital, South Brisbane, Queensland
  - Mercy Hospital for Women, Heidelberg, Victoria
  - King Edward Memorial Hospital, Perth, Western Australia
- Canada (2):
  - Fraser Health Surrey Memorial Hospital, Surrey, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- University of Cologne, Cologne, Germany
- Japan (6):
  - Kyorin University Hospital, Shinkawa, Mitaka
  - Nagano Children's Hospital, Azumino, Nagano
  - Osaka Women's & Children's Hospital, Izumi, Osaka
  - Saitama Medical Center, Saitama Medical University, Kawagoe, Saitama
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - National Center for Child Health and Development, Tokyo
- La Paz Hospital, La Paz, Spain
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Background] Rysavy M, Nakamura T, Mehler K, Agren J, McNamara P, Backes C; Tiny Baby Collaborative. Use of 2.0-mm endotracheal tubes for periviable infants. J Perinatol. 2022 Sep;42(9):1275-1276. doi: 10.1038/s41372-022-01323-7. Epub 2022 Jan 26. No abstract available. PMID 35082430
- [Background] Rysavy MA, Mehler K, Oberthur A, Agren J, Kusuda S, McNamara PJ, Giesinger RE, Kribs A, Normann E, Carlson SJ, Klein JM, Backes CH, Bell EF. An Immature Science: Intensive Care for Infants Born at </=23 Weeks of Gestation. J Pediatr. 2021 Jun;233:16-25.e1. doi: 10.1016/j.jpeds.2021.03.006. Epub 2021 Mar 7. No abstract available. PMID 33691163
- See also: Related Info — https://www.tinybabycollaborative.org